CLINICAL TRIAL: NCT03910127
Title: A Phase Ib, Multicenter, Randomized Study to Evaluate the Pharmacokinetics, Efficacy and Safety of TQB2450 Combined With or Without Anlotinib in Patients With Advanced Non-small Cell Lung Cancer（NSCLC）
Brief Title: Study of TQB2450 Combined With Anlotinib in Patients With Advanced Non-small Cell Lung Cancer（NSCLC）
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TQB2450-Ib-01
Record Dates: First submitted 2019-04-02; First posted 2019-04-10 (Actual); Last update posted 2019-10-30 (Actual); Status verified 2019-01

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — anlotinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- TQB2450 + Anlotinib (10 mg) (Experimental): TQB2450 1200 mg administered intravenously (IV) on Day 1 of each 21-day cycle plus Anlotinib capsules 10 mg given orally in fasting conditions, once daily in 21-day cycle (14 days on treatment from Day 1-14, 7 days off treatment from Day 15-21)
  Interventions: Drug: TQB2450; Drug: Anlotinib
- TQB2450 + Anlotinib (12 mg) (Experimental): TQB2450 1200 mg administered IV on Day 1 of each 21-day cycle plus Anlotinib capsules 12 mg given orally in fasting conditions, once daily in 21-day cycle (14 days on treatment from Day 1-14, 7 days off treatment from Day 15-21)
  Interventions: Drug: TQB2450; Drug: Anlotinib
- TQB2450 + Placebo (Placebo Comparator): TQB2450 1200 mg administered IV on Day 1 of each 21-day cycle plus Placebo for Anlotinib capsules given orally in fasting conditions, once daily in 21-day cycle (14 days on treatment from Day 1-14, 7 days off treatment from Day 15-21)
  Interventions: Drug: TQB2450; Drug: Anlotinib

INTERVENTIONS:
Drug: TQB2450 — TQB2450 is a humanized monoclonal antibody targeting programmed death ligand-1 (PD-L1), which prevents PD-L1 from binding to PD-1 and B7.1 receptors on T cell surface, restores T cell activity, thus enhancing immune response and has potential to treat various types of tumors.
Drug: Anlotinib — a multi-target receptor tyrosine kinase inhibitor
  Arms: TQB2450 + Anlotinib (10 mg); TQB2450 + Anlotinib (12 mg)
Drug: Anlotinib — matching placebo
  Arms: TQB2450 + Placebo

SUMMARY:
TQB2450 is a humanized monoclonal antibody targeting programmed death ligand-1 (PD-L1), which prevents PD-L1 from binding to PD-1 and B7.1 receptors on T cell surface, restores T cell activity, thus enhancing immune response and has potential to treat various types of tumors.

ELIGIBILITY:
Inclusion Criteria:

1.18 years and older; Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1; Life expectancy ≥ 3 months.

2. Histologically or cytologically confirmed Epidermal Growth Factor Receptor (EGFR)/ Anaplastic Lymphoma Kinase (ALK) wild type non-small cell lung cancer.

3. Advanced patients who had received at least first-line of standard chemotherapy but failed or intolerable , with at least one measurable lesion based on RECIST 1.1.

4. PD-L1-positive tumor status (TPS≥1%) as determined by an immunohistochemistry (IHC) assay based on PD-L1 expression on tumor infiltrating immune cells and/or tumor cells performed by a central laboratory.

5.The main organs function are normally, the following criteria are met:

1. routine blood tests：hemoglobin (Hb)≥90g/L (no blood transfusion and blood products within 14 days); absolute neutrophil count (ANC) ≥1.5×109/L; platelets (PLT) ≥80×109/L;
2. Blood biochemical examination: alanine transaminase (ALT) and aspartate aminotransferase (AST)≤ 2.5×ULN (when the liver is invaded，≤ 5×ULN);total bilirubin (TBIL)≤1.5×ULN (Gilbert syndrome patients，≤ 3×ULN)；serum creatinine (Cr) ≤1.5×ULN，or calculated creatinine clearance (CrCl) ≥50ml/min； calculated creatinine clearance formula：Ccr=(140-age)×weight(kg)/72×Scr(mg/dl) Ccr=[(140-age)×weight(kg)]/[0.818×Scr(umol/L) (According to the calculation results , female Patients ×0.85；1 mg/dL = 88.41 umol/ L)
3. Coagulation function: activated partial thromboplastin time (aPTT) ,international normalized ratio (INR) ,prothrombin time (PT) ≤1.5×ULN；
4. left ventricular ejection fraction (LVEF) measured by the Cardiac echocardiography ≥ 50%.

   6. Male or female subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 6 months after the last dose of study (such as intrauterine devices , contraceptives or condoms) ；No pregnant or breastfeeding women, and a negative pregnancy test are received within 7 days before the randomization.

   7. Understood and signed an informed consent form.

Exclusion Criteria:

1. Prior therapy with Anlotinib, anti-programmed cell death (PD)-1, anti-PD-L1 or other immunotherapy against PD-1/PD-L1.
2. Severe hypersensitivity occurs after administration of other monoclonal antibodies.
3. Diagnosed and/or treated additional malignancy within 5 years prior to randomization with the exception of cured basal cell carcinoma of skin and carcinoma in situ of cervix.
4. Has any active autoimmune disease or history of autoimmune disease, such as autoimmune hepatitis, interstitial pneumonia, enteritis, vasculitis, nephritis, asthma patients who need bronchiectasis for medical intervention; Subjects with the vitiligo without systemic treatment, psoriasis, alopecia, well-controlled type I diabetes mellitus, hypothyroidism stable on hormone replacement will not be excluded from this study.
5. Immunosuppressive therapy with immunosuppressive agents or systemic or absorbable local hormones (dosage > 10 mg/day prednisone or other therapeutic hormones) is required for the purpose of immunosuppression.
6. Has multiple factors affecting oral medication, such as inability to swallow, post-gastrointestinal resection, chronic diarrhea and intestinal obstruction, etc.
7. Has uncontrollable pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures.
8. Imaging (CT or MRI) shows that tumor invades large blood vessels or the boundary with blood vessels is unclear.
9. Has any bleeding or bleeding events ≥ grade 3 or with unhealed wounds, ulcerative , or fractures within 4 weeks prior to the first administration.
10. Has uncontrollable symptoms of brain metastases, spinal cord compression, cancerous meningitis within 8 weeks before the first-dosing, or brain or leptomeningeal disease found by CT or MRI during screening.
11. Has received chemotherapy, surgery, radiotherapy, the last treatment from the first dose less than 4 weeks, or oral targeted drugs for less than 5 half-lives, or oral fluorouracil pyridine drugs for less than 14 days, mitomycin C and nitrosourea for less than 6 weeks. Patients whose adverse events (except alopecia) caused by previous treatment did not recover to ≤ grade 1.
12. Patients with any serious and/or uncontrollable disease, including :

    1. Has poor blood pressure control, systolic blood pressure ≥ 150 mmHg, diastolic blood pressure ≥ 90 mmHg;
    2. Thrombotic events, ischemic attacks, myocardial infarction, grade 2 congestive heart failure or arrhythmias requiring treatment including QTc ≥ 480ms occurred within 6 months of first administration;
    3. Severe active or uncontrolled infections ≥ grade 2;
    4. Has known clinical history of liver diseases, including viral hepatitis, known carriers of hepatitis B virus (HBV) must exclude active HBV infection, that is, HBV DNA positive > 1 *104 copies/mL or > 2000 IU/mL, known hepatitis C virus infection (HCV) and HCV RNA positive > 1 *103 copies/mL, or other decompensated hepatitis and chronic hepatitis, which require antiviral treatment;
    5. HIV positive;
    6. Poor control of diabetes mellitus, fasting blood-glucose ≥ grade 2;
13. Has vaccinated with vaccines or attenuated vaccines within 4 weeks prior to first administration.
14. According to the judgement of the researchers, there are other factors that may lead to the termination of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2019-06-11 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | up to approximately 18 months
  PFS defined as the time from randomization until the first documented progressive disease (PD) or death from any cause.

SECONDARY OUTCOMES:
Adverse Event （AE）: Drug dose adjustment | up to approximately 18 months
  Security Index
Overall response rate （ORR） | up to approximately 18 months
  Percentage of Participants Achieving Complete Response (CR) and Partial Response (PR)
Disease control rate（DCR） | up to approximately 18 months
  Percentage of Participants Achieving Complete Response (CR) and Partial Response (PR) and Stable Disease (SD).
Overall survival (OS) | up to approximately 24 months
  OS defined as the time from randomization to death from any cause. Participants who do not die at the end of the extended follow-up period, or were lost to follow-up during the study, were censored at the last date they were known to be alive.
Pharmacokinetics (PK): Maximum Concentration (Cmax) | Hour 0 (before infusion), 30 minutes after start of infusion, 0, 2, 6, 10, 24, 72, 168, 336, 504 hours after end of infusion on cycle 1 and cycle 6 (each cycle is 21 days).
  The Cmax is observed maximum serum concentration, taken directly from the serum concentration-time profile
Pharmacokinetics (PK): Area Under the Serum Concentration-Time Curve From Time Zero to Infinite Time (AUC[0-infinity]) | Hour 0 (before infusion), 30 minutes after start of infusion, 0, 2, 6, 10, 24, 72, 168, 336, 504 hours after end of infusion on cycle 1 and cycle 6 (each cycle is 21 days).
  The AUC(0-infinity) is area under the serum concentration-time curve from time zero to infinite time.
Pharmacokinetics (PK): t1/2 | Hour 0 (before infusion), 30 minutes after start of infusion, 0, 2, 6, 10, 24, 72, 168, 336, 504 hours after end of infusion on cycle 1 and cycle 6 (each cycle is 21 days).
  Terminal half-life

CONTACTS AND LOCATIONS:
Overall Officials: Baohui Han, Doctor, Principal Investigator — Shanghai Chest Hospital; Kai Li, Doctor, Principal Investigator — Tianjin Cancer Hospital
Locations (3):
- China (3):
  - Gansu Province Tumor Hospital, Lanzhou, Gansu
  - Henan Province Tumor Hospital, Luoyan, Henan
  - Jilin Cancer Hospital, Changchun, Jilin